CLINICAL TRIAL: NCT05168852
Title: Evaluation of Clinical Performance of Permanent Resin Restorations Fabricated by 3D Printer
Brief Title: Permanent Resin Restorations Fabricated by Three Dimension Printer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, zeliha gonca bek kurklu, department of dentistry, Cukurova University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: cu scientific research unit
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Three-Dimensional Printing, Computer-Aided Design, Dental

STUDY DESIGN:
Intervention Model Description: After the restorations are applied, the patients are checked in the 1st week and 6th months.
Who Masked: Participant
Masking Description: Individuals aged 18-65 years with a D1 or D2 class II carious lesion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Permanent Resin 1 week (Experimental): 1st week control
  Interventions: Other: Formlabs Permanent CB Resin
- Permanent Resin 6 mouth (Experimental): 6th month control
  Interventions: Other: Formlabs Permanent CB Resin

INTERVENTIONS:
Other: Formlabs Permanent CB Resin — Tooth-colored, ceramic-filled permanent resin that can be fabricated with a 3D printer

SUMMARY:
Additive manufacturing (AM) and 3D printing (3DP) technologies have advanced significantly in many different areas. With the time and cost advantage it provides in low-volume production, 3D printing technologies also come to the fore in the field of digital dentistry. A tooth-coloured, ceramic-filled permanent resin has been introduced by the manufacturer for the 3D fabrication of permanent single crowns, veneers, inlays and onlays. The aim of this clinical study was to clinically evaluate the long-term survival and intraoral performance of 3D-printed permanent resin. to the ICDAS caries classification system, 20 volunteers between the ages of 18-65 with class II caries lesion at D1 or D2 level were included in this study. Restorations were checked 1 week (baseline) and 6 months after completion and scored using the Modified Ryge Criteria (USPHS2(United States Public Health Service)). Statistical analysis was done by Kaplan-Meier survival analysis.

DETAILED DESCRIPTION:
The design and manufacture of 3D printed restorations relies on the exchange of digital information (data) between 3D imaging, 3D virtual planning and/or 3D printing technologies. One of the key points in the widespread use of 3D printers is the emergence of these systems that allow data from different sources to be used in a personal computer with various design and production technologies. It saves Digital Imaging and Communication in Medicine (DICOM) files in STL format. STL files can be printed and processed with various CAD/CAM systems in local manufacturing or remote labs. This is an important advantage of using open source. With these systems, it is possible to produce restorations with clearer anatomical features thanks to current 3D printing technologies. In other words, low-cost restorations with more useful properties can be produced.

ELIGIBILITY:
Inclusion Criteria:

* premolar and/or molar tooth has class II caries lesion at D1 or D2 level according to ICDAS caries classification system.

Exclusion Criteria:

* bad oral hygiene
* bruxism,
* malocclusion,
* dry mouth,
* periodontal disease,
* teeth with restoration,
* periodontal or periapical pathology non-opposite and/or non-contact teeth will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
1 week follow up | 1 week
  Restorations will be scored 1 week after it is cemented onto the tooth using the Modified Ryge Criteria (USPHS2(United States Public Health Services))

SECONDARY OUTCOMES:
6 mouths follow up | 6 mouths
  Restorations will be scored 6 mouths after it is cemented onto the tooth using the Modified Ryge Criteria (USPHS2(United States Public Health Services))

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Faculty of Dentistry, Department of Restorative Dentistry, Adana, Sarıcam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No